Single-used versus MultiPIE-used endotracheal suCtIon cAtheters in mechanically ventiLated ICU patients: the SPECIAL-ICU trial. Informed consent form Version 1 dated 14<sup>th</sup> of December 2023.

## Single-used versus MultiPIE-used endotracheal suCtion cAtheters in mechanically ventiLated ICU patients: the SPECIAL-ICU trial

**Short title: SPECIAL-ICU trial** 

**Informed Consent Form, Version 1** 

Dated 14th of December 2023

Single-used versus MultiPIE-used endotracheal suCtIon cAtheters in mechanically ventiLated ICU patients: the SPECIAL-ICU trial. Informed consent form Version 1 dated 14<sup>th</sup> of December 2023.

## Appendix III: Informed consent form (ICF) for patient participation

## **Participant Study Number**

## **CONSENT FORM**

Title of the Project: Single-used versus MultiPIE-used endotracheal suCtion cAtheters in mechanically ventiLated ICU patients: the SPECIAL-ICU trial

Name of Researcher: Mr Mohamed H. Eid (PhD Student)

| | | | PI | ease initial box |
|---|---|---|---|---|
| 1. | I confirm that I have read and under <b>December 2023 (version 1.0)</b> for the consider the information, ask questions satisfactorily. | | | |
| 2. | I understand that my relative participation is voluntary and that I am free to withdraw him/her at any time, without giving any reason, without his/her medical care or legal rights being affected. | | | |
| 3. | I understand that relevant sections of any of my relative's medical notes and data collected during the study may be looked at by responsible individuals from the University of Plymouth, or the regulatory authorities, where it is relevant to my relative taking part in this research. I give permission for these individuals to have access to my relative's records. | | | |
| 4. | I agree that information collected about my relative during the course of the study will be stored confidentially and securely on University of Plymouth premises in accordance with the Data Protection Act 1998. | | | |
| 5. | I agree to my intensive care unit relative's participation in the study. | | | |
| 6. | I agree to allow my relative to take part in the above study. | | | |
| Name of participant | | Date | Signature | <u> </u> |
| Name of person taking consent | | <br>Date | Signature | <br>Signature |

When completed: 1 for participant; 1 for researcher site file; 1 to be kept in medical notes.